CLINICAL TRIAL: NCT06620211
Title: Evaluation of the Safety, Performance, and Tolerability of the Sacromesh® Medical Device in the Treatment of Prolapse by Promontofixation in a Population of Patients Followed Over the Long Term.
Acronym: SCUPP
Status: Completed | Type: Observational
Sponsor: Cousin Biotech (Industry)
Responsible Party: Sponsor
Other Study IDs: RC-P-T3-33
Record Dates: First submitted 2023-12-08; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Prolapse; Female
MeSH Terms: conditions — Prolapse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: promontofixation, prolapse cure — Patient who underwent surgery to place the Sacromesh® medical device (promontofixation) for a prolapse cure, between 2009 and 2018

SUMMARY:
An observational, multicenter study with retrospective recruitment and two data collection methods, one retrospective (medical records) and the other prospective (questionnaires).

Patients who meet the inclusion criteria and have none of the non-inclusion criteria will be selected using the computer database of each investigating center. Data from consultation visits and surgery data will be collected and filled in the observation books.

The patient will be contacted by the investigators to collect data on quality of life and the existence or absence of pain associated with implant placement at follow-up.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for participation in the study are as follows:

• Patient who underwent surgery to place the Sacromesh® medical device for a prolapse cure, between 2009 and 2018 in one of the investigation centres participating in the study.

• Patient who has read the information note and has not formulated an -opposition.

• Adult patient with full mental capacity/capability

Exclusion Criteria:

• Patient under guardianship or curatorship

• Patient hospitalized at time of inclusion

• Patient with an adjacent pathology that may strongly interfere with her quality of life and VAS score.

* Patients with mental psychological pathology

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prolapse cure, female only
Study Population: SCUPP is an observational retrospective study without any planed comparison. This is a multicentric study and from the center with the best recruitment potential, 5 centers were selected.
  The primary endpoint is the rate of reoperation which is expected to be very small according to previous investigation for Sacromesh® and according to literature. For example, a study investigated perioperative and mid-term clinical outcomes after laparoscopic sacrocolpopexy (LSCP) with light titanium-coated polypropylene (TCP) mesh in a large group of patients affected by International Continence Society stage II-IV pelvic organ prolapse (POP) reported a posterior recurrence of about 0.4% (1 out of 217 patients) [Campagna et al., 2020]. Another study investigating the Robotic sacrocolpopexy (RSCP) option for the treatment of apical, anterior, and proximal posterior compartment pelvic organ prolapses reported a POP recurrence of about 2% (2 out of 91 patients) [Li Marzi et al., 2022].
Sampling Method: Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
RATE AND TYPE OF REINTERVENTION | 2020 - 2023
  safety assessment of Sacromesh® implan through the documentation, within the French healthcare context, of the rate and type of re-interventions after Sacromesh® implantation. Collection and documentation of the nature and frequency of reinterventions after placement of the Sacromesh® device, including causes and nature of eventual explants, be it total or partial. The rate of re intervention will be calculated using Yes/No answer to POP recurrence question in the CRF. Yes answer to the question will be considered as a re intervention. In case of any POP recurrence investigator was asked to fill an adverse event form to describe the re intervention. Type of re intervention will be derived from AE form into a two classes categorical variable taking either 'De novo prolapse (recurrence, vaginal extrusion)' or 'Other' value. Both rate of re intervention and type of re intervention will be described as qualitative variables.

SECONDARY OUTCOMES:
evaluation the tolerance of the Sacromesh® implant Rate and type of postoperative complications | 2020 - 2023
  Rate and type of postoperative complications The rate and type of postoperative complications will be presented as mean (standard deviation [SD]), median, 1st and 3rd quartiles, range, and the 95% (CI) based on the Student-t distribution.
evaluation the tolerance of the Sacromesh® implant qol | 2020 - 2023
  Quality of life Two questionnaires will be assessed: PFIQ-7 and PFDI-20 questionnaires. Results will be presented as mean (standard deviation [SD]), median, 1st and 3rd quartiles, range, and the 95% (CI) based on the Student-t distribution. All applicable statistical tests will be two-sided and will be performed using a 5% significance level; CI presented will be 95%.
evaluation the tolerance of the Sacromesh® implant postoperative pain | 2020 - 2023
  Postoperative pain Pain will be assessed with VAS scale and expressed as a mean (standard deviation [SD]), median, 1st and 3rd quartiles, range, and the 95% (CI) based on the Student-t distribution. All applicable statistical tests will be two-sided and will be performed using a 5% significance level; CI presented will be 95%.

CONTACTS AND LOCATIONS:
Locations (1):
- Cousin Biotech, Wervicq-Sud, France

IPD SHARING:
Plan to Share IPD: Undecided